CLINICAL TRIAL: NCT00541229
Title: A Phase 1b, Multicenter, Double-Blind, Randomized, Placebo-Controlled, Crossover Clinical Trial of Sitagliptin 100 mg and Sitagliptin 200 mg in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Diet and Exercise
Brief Title: Sitagliptin Dose Comparison Study in Patients With Type 2 Diabetes (MK-0431-077)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-077; 2007_533
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Results first posted 2009-07-28 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): sitagliptin 100 mg
  Interventions: Drug: sitagliptin phosphate
- 2 (Experimental): sitagliptin 200 mg
  Interventions: Drug: sitagliptin phosphate
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: sitagliptin phosphate — sitagliptin 100 mg tablets q.d. (once daily) for 7 days.
  Other Names: MK0431
  Arms: 1
Drug: sitagliptin phosphate — sitagliptin 200 mg tablets q.d. (once daily) for 7 days.
  Other Names: MK0431
  Arms: 2
Drug: Comparator: Placebo — sitagliptin 100 mg & 200 mg matching Placebo tablets q.d. (once daily) for 7 days.
  Arms: 3

SUMMARY:
A study to assess the safety and efficacy of sitagliptin 100mg compared to sitagliptin 200mg in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patient has Type 2 Diabetes
* Patient is between the ages of 30-65 years
* Patient is not on an antihyperglycemic agent (AHA) (glycosylated hemoglobin [A1C] 7-10% ), or is on oral single AHA or low-dose combination therapy (A1C 6.5-9.5%).

Exclusion Criteria:

* Patient has Type 1 Diabetes
* Patient has been treated with sitagliptin, vildagliptin, or other similar drugs or has been treated with exenatide in the past 3 months
* Patient has taken insulin within the past 3 months

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-08-24 (Actual); Primary Completion 2008-06-17 (Actual); Study Completion 2008-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Alba M, Sheng D, Guan Y, Williams-Herman D, Larson P, Sachs JR, Thornberry N, Herman G, Kaufman KD, Goldstein BJ. Sitagliptin 100 mg daily effect on DPP-4 inhibition and compound-specific glycemic improvement. Curr Med Res Opin. 2009 Oct;25(10):2507-14. doi: 10.1185/03007990903209514. PMID 19691426

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 17-Oct-2007; Last Patient Last Visit: 01-Jul-2008; Seventeen medical clinics worldwide (8 in the United States, 8 in Europe and 1 in Mexico).
Pre-assignment Details: Following a 4-week (wk) diet/exercise (and wash-off period for patients on antihyperglycemic agent [AHA]), patients with fasting plasma glucose (FPG) 130-250 mg/dL were eligible to enter a 2-wk placebo run-in period prior to randomization.
Groups:
- Placebo / 100 mg / 200 mg: Placebo / 100 mg / 200 mg Group includes patients receiving once daily administration of the following treatments: sitagliptin-matching placebo in Treatment Period I, sitagliptin 100 mg in Treatment Period II (after Washout Period I), and sitagliptin 200 mg in Treatment Period III (after Washout Period II)
- 100 mg / 200 mg / Placebo: 100 mg / 200 mg / Placebo Group includes patients receiving once daily administration of the following treatments: sitagliptin 100 mg in Treatment Period I, sitagliptin 200 mg in Treatment Period II (after Washout Period I), and sitagliptin-matching placebo in Treatment Period III (after Washout Period II)
- 200 mg / Placebo / 100 mg: 200 mg / Placebo / 100 mg Group includes patients receiving once daily administration of the following treatments: sitagliptin 200 mg in Treatment Period I, sitagliptin-matching placebo in Treatment Period II (after Washout Period I), and sitagliptin 100 mg in Treatment Period III (after Washout Period II)
- Placebo / 200 mg / 100 mg: Placebo / 200 mg / 100 mg Group includes patients receiving once daily administration of the following treatments: sitagliptin-matching placebo in Treatment Period I, sitagliptin 200 mg in Treatment Period II (after Washout Period I), and sitagliptin 100 mg in Treatment Period III (after Washout Period II)
- 100 mg / Placebo / 200 mg: 100 mg / Placebo / 200 mg Group includes patients receiving once daily administration of the following treatments: sitagliptin 100 mg in Treatment Period I, sitagliptin-matching placebo in Treatment Period II (after Washout Period I), and sitagliptin 200 mg in Treatment Period III (after Washout Period II)
- 200 mg / 100 mg / Placebo: 200 mg / 100 mg / Placebo includes patients receiving once daily administration of the following treatments: sitagliptin 200 mg in Treatment Period I, sitagliptin 100 mg in Treatment Period II (after Washout Period I), and sitagliptin-matching placebo in Treatment Period III (after Washout Period II)
Period: Treatment Period I (Week 1)
Arm/Group | Placebo / 100 mg / 200 mg | 100 mg / 200 mg / Placebo | 200 mg / Placebo / 100 mg | Placebo / 200 mg / 100 mg | 100 mg / Placebo / 200 mg | 200 mg / 100 mg / Placebo
Started | 17 | 16 | 20 | 18 | 14 | 18
Completed | 17 | 15 | 17 | 17 | 14 | 16
Not Completed | 0 | 1 | 3 | 1 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Specified Criteria | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 1 | 2 | 1 | 0 | 0
Period: Washout Period I (Week 2-5)
Arm/Group | Placebo / 100 mg / 200 mg | 100 mg / 200 mg / Placebo | 200 mg / Placebo / 100 mg | Placebo / 200 mg / 100 mg | 100 mg / Placebo / 200 mg | 200 mg / 100 mg / Placebo
Started | 17 | 15 | 17 | 17 | 14 | 16
Completed | 13 | 13 | 13 | 13 | 13 | 11
Not Completed | 4 | 2 | 4 | 4 | 1 | 5
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 3 | 2 | 3 | 3 | 1 | 4
Period: Treatment Period II (Week 6)
Arm/Group | Placebo / 100 mg / 200 mg | 100 mg / 200 mg / Placebo | 200 mg / Placebo / 100 mg | Placebo / 200 mg / 100 mg | 100 mg / Placebo / 200 mg | 200 mg / 100 mg / Placebo
Started | 13 | 13 | 13 | 13 | 13 | 11
Completed | 11 | 12 | 12 | 12 | 11 | 8
Not Completed | 2 | 1 | 1 | 1 | 2 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Study Terminated by Sponsor | 2 | 1 | 1 | 1 | 1 | 2
Period: Washout Period II (Week 7-10)
Arm/Group | Placebo / 100 mg / 200 mg | 100 mg / 200 mg / Placebo | 200 mg / Placebo / 100 mg | Placebo / 200 mg / 100 mg | 100 mg / Placebo / 200 mg | 200 mg / 100 mg / Placebo
Started | 11 | 12 | 12 | 12 | 11 | 8
Completed | 7 | 8 | 10 | 8 | 7 | 5
Not Completed | 4 | 4 | 2 | 4 | 4 | 3
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 3 | 4 | 2 | 4 | 3 | 3
Period: Treatment Period III (Week 11)
Arm/Group | Placebo / 100 mg / 200 mg | 100 mg / 200 mg / Placebo | 200 mg / Placebo / 100 mg | Placebo / 200 mg / 100 mg | 100 mg / Placebo / 200 mg | 200 mg / 100 mg / Placebo
Started | 7 | 8 | 10 | 8 | 7 | 5
Completed | 7 | 8 | 9 | 8 | 6 | 4
Not Completed | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Specified Criteria | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo / 100 mg / 200 mg | 100 mg / 200 mg / Placebo | 200 mg / Placebo / 100 mg | Placebo / 200 mg / 100 mg | 100 mg / Placebo / 200 mg | 200 mg / 100 mg / Placebo | Total
Number analyzed (Participants) | 17 | 16 | 20 | 18 | 14 | 18 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (8.4) | 56.6 (5.8) | 55.7 (7.2) | 55.3 (8.3) | 50.0 (10.0) | 48.6 (9.6) | 53.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 7 | 4 | 4 | 3 | 28
  Male | 12 | 11 | 13 | 14 | 10 | 15 | 75
Race/Ethnicity, Customized [Number; unit: participants]
  White | 12 | 14 | 15 | 15 | 11 | 12 | 79
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Other | 5 | 2 | 5 | 3 | 3 | 5 | 23
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 179.3 (32.1) | 167.0 (41.1) | 184.0 (42.1) | 173.2 (43.2) | 158.5 (17.3) | 166.0 (36.5) | 172.0 (36.9)

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Weighted Mean Glucose (WMG)
Description: The 24-hour WMG was calculated as the area under the 24-hour glucose curve (AUC(0-24 hr)) divided by 24 using linear trapezoidal method.
Time Frame: Day 7 of Treatment Period I. Due to a carry-over effect that was observed between treatment periods, efficacy results are presented from Treatment Period I only.
Population: The per-protocol (PP) population consisted of all patients randomized who had a measurement at Day 7 in Treatment Period I and did not have any major protocol violations. Missing data were not imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Groups:
- Sitagliptin 200mg: Sitagliptin 200 mg group included the Treatment Period I data from patients randomized to treatment sequence Sitagliptin 200 mg/Sitagliptin 100 mg/placebo and treatment sequence Sitagliptin 200 mg/ placebo/ Sitagliptin 100 mg.
- Sitagliptin 100mg: Sitagliptin 100 mg group included the Treatment Period I data from patients randomized to treatment sequence Sitagliptin 100 mg/Sitagliptin 200 mg/placebo and treatment sequence Sitagliptin 100 mg/ placebo/ Sitagliptin 200 mg.
- Placebo: Placebo group included the Treatment Period I data from patients randomized to treatment sequence placebo/Sitagliptin 100 mg/Sitagliptin 200 mg and treatment sequence placebo/Sitagliptin 200 mg/Sitagliptin 100 mg.
Arm/Group | Sitagliptin 200mg | Sitagliptin 100mg | Placebo
Number analyzed (Participants) | 28 | 26 | 30
mg/dL | 169.1 [153.8 to 184.4] | 159.0 [143.1 to 174.9] | 200.9 [186.1 to 215.7]
Statistical Analysis 1: Comparison: Sitagliptin 200mg vs Placebo; For this comparison, the mean in the placebo group was subtracted from the mean in the sitagliptin 200 mg group; Test type: Superiority or Other; p = 0.004, ANOVA; Model term: treatment; Mean Difference (Final Values) = -31.8, 95% CI [-53.1 to -10.5]
Statistical Analysis 2: Comparison: Sitagliptin 100mg vs Placebo; For this comparison, the mean in the placebo group was subtracted from the mean in the sitagliptin 100 mg group; Test type: Superiority or Other; p < 0.001, ANOVA; Model term: treatment; Mean Difference (Final Values) = -41.9, 95% CI [-63.6 to -20.2]
Statistical Analysis 3: Comparison: Sitagliptin 200mg vs Sitagliptin 100mg; This was pre-defined as a non-superiority test, i.e., to show that sitagliptin 200 mg is not superior to sitagliptin 100 mg. For this comparison, the mean in the sitagliptin 100 mg group was subtracted from the mean in the sitagliptin 200 mg group; Test type: Non-Inferiority or Equivalence — The hypothesis stated that the lower bound of 80% one-sided confidence interval for the comparison in 24-hour WMG reduction between sitagliptin 200 mg and sitagliptin 100 mg is above -5 mg/dL; Mean Difference (Final Values) = 10.1, 80% CI [0.61 to 9999999] — This is a 1-sided 80% confidence interval and the upper bound 9999999 was used here to indicate positive infinity

ADVERSE EVENTS:
Groups:
- Sitagliptin 200 mg: Sitagliptin 200 mg Group included data from all randomized patients in treatment periods with once-daily administration of sitagliptin 200 mg. Due to the crossover design, patients are counted in the denominator for each treatment that they received. Patients are counted in the numerator for the treatment that they were receiving at the time when the AE occurred.
- Sitagliptin 100 mg: Sitagliptin 100 mg Group included data from all randomized patients in treatment periods with once-daily administration of sitagliptin 100 mg. Due to the crossover design, patients are counted in the denominator for each treatment that they received. Patients are counted in the numerator for the treatment that they were receiving at the time when the AE occurred.
- Placebo: Placebo Group included data from all randomized patients in treatment periods with once-daily administration of sitagliptin-matching placebo tablets. Due to the crossover design, patients are counted in the denominator for each treatment that they received. Patients are counted in the numerator for the treatment that they were receiving at the time when the AE occurred.
Arm/Group | Sitagliptin 200 mg | Sitagliptin 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/72 | 0/74
Other Adverse Events (participants affected / at risk) | 4/78 | 2/72 | 4/74
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin 200 mg (N=78) | Sitagliptin 100 mg (N=72) | Placebo (N=74)
Headache (Nervous system disorders) | 4 | 2 | 4

LIMITATIONS AND CAVEATS:
The pre-specified rule for non-superiority of sitagliptin 200 mg compared with 100 mg was met at the planned interim analysis. As such, the trial was terminated as pre-specified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.